CLINICAL TRIAL: NCT06573801
Title: A Single Centre Randomised Prospective Cross-over Study to Assess Agreement Between Blood Pressure Measurements Taken Using Cuffless Wearable and Cuffed, Ambulatory Blood Pressure Monitoring Devices.
Brief Title: Comparing Accuracy Between Cuffless Wrist Worn and Cuffed Ambulatory BP Monitoring Devices
Acronym: Continuum BP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 341847
Record Dates: First submitted 2024-08-13; First posted 2024-08-27 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Blood Pressure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aktiia (Active Comparator): Participants will wear the Aktiia Bracelet for 24h alongside a cuffed ambulatory BP monitor. Both devices will be recording BP at pre programmed intervals.
  Interventions: Device: Aktiia Bracelet; Device: Spacelabs OnTrak Ambulatory Blood Pressure monitor
- Healthstats (Active Comparator): Participants will wear the Healthstats BPro Evo smart watch for 24h alongside a cuffed ambulatory BP monitor. Both devices will be recording BP at pre programmed interval
  Interventions: Device: Healthstats BPro Evo; Device: Spacelabs OnTrak Ambulatory Blood Pressure monitor

INTERVENTIONS:
Device: Aktiia Bracelet — Wrist worn bracelet with an optical sensor that measures pulse wave characteristics at the wrist.
  Arms: Aktiia
Device: Healthstats BPro Evo — Wrist worn watch that uses applanation tonometry to measure pulse wave characteristics at the wrist.
  Arms: Healthstats
Device: Spacelabs OnTrak Ambulatory Blood Pressure monitor — Cuffed ambulatory BP monitor that will measure upper arm BP using oscillometry.

SUMMARY:
Wrist worn devices can help record Blood Pressure (BP) throughout the day. As such devices are becoming increasingly affordable, they could help improve awareness, early diagnosis, and treatment of high and uncontrolled BP.

The goal of Continuum BP is to evaluate how BP readings from two different types of wrist-worn cuffless devices available on the market (Aktiia and Healthstats BPro Evo) compare with BP taken using an ambulatory BP monitor which records readings over 24h using a standard upper arm cuff. This interventional study will recruit balanced numbers of male and female participants within different age group, who will sequentially wear the Aktiia Bracelet and the Heathstats BPro Evo for a period of 24h, alongside the cuffed ambulatory BP monitor.

If wrist worn devices are found to measure BP reliably, future research will assess if artificial intelligence can use continuous BP readings from these devices to learn patterns and changes in BP; and develop digital twin models to guide better, more precise BP management for individuals.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is aged ≥21 years and <85 years at the time of screening visit.
2. Able to speak and understand English.
3. Able and willing to give informed consent.
4. Independent and mobile.
5. Willing and able to wear devices/no upper limb restrictions.

Exclusion Criteria:

1. Individuals who are or have been involved in interventional research within a period of 3 months.
2. Vulnerable individuals including those with mental ill-health or who are care dependant.
3. Individuals with serious comorbidities or end organ damage (e.g., previously diagnosed heart failure with New York Heart Association class III/IV, verbal or documented evidence of renal failure or history of dialysis, stroke or myocardial infarction within the last 1-year, previous stroke with residual deficit); and doctor diagnosed hyperthyroidism.
4. Individuals with arterio-venous fistula; or reduced peripheral perfusion identified by a history of Raynaud's syndrome or a pulse pressure of <30mmHg or a capillary refill time of >3s in the dominant arm.
5. Individuals with heart rhythm disorders e.g., persistent Atrial Fibrillation and those who have tachycardia > 120 after 5 minutes of rest.
6. Individuals with skin irritation injury or damage.
7. Self-reported pregnancy. Participation will be withdrawn in the event of pregnancy following enrolment.
8. Life threatening or terminal illness with limited lifespan of <12months.
9. Obesity (Body Mass Index 35kg/m2 or higher) or arm/wrist circumferences outside the range highlighted in each device's specification.
10. Those with very high office BP (greater than Stage 3 hypertension).
11. Interarm difference >15mmHg in Systolic BP and >10mmHg in Diastolic BP.
12. Where the PI thinks that it would be technically difficult to obtain or interpret blood pressures measurements.

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2025-01-28 (Actual); Primary Completion 2025-11-19 (Actual); Study Completion 2025-11-19 (Actual)

PRIMARY OUTCOMES:
Mean Daytime BP Difference | Up to 24 hours from device application, using readings from 7am to 11pm.
  Difference in average Systolic and Diastolic BP measured using ambulatory BP monitor and each device over daytime.

SECONDARY OUTCOMES:
Mean 24 hours BP Difference | Up to 24 hours from device application.
  Difference in average Systolic and Diastolic BP measured using ambulatory BP monitor and each device over 24 hours.
Mean Nighttime BP Difference | Up to 24 hours from device application, using readings from 11pm to 7am.
  Difference in average Systolic and Diastolic BP measured using ambulatory BP monitor and each device over night-time.
Difference in Blood Pressure Variability | Up to 24 hours from device application, using readings from 7am to 11pm to indicate daytime and 11pm to 7am to indicate night-time.
  Difference in BP variability during daytime and night-time BP recorded by ambulatory BP monitor and each device.
Acceptability of wearing cuffless BP devices using a (simple non-validated) Likert-type device wearability questionnaire. | Up to 24 hours from device application
  Measure(s) of acceptability of wearing cuffless BP monitors (compared with wearing ambulatory BP monitor) will include comfort, ability to carry on daily activities, interference with sleep and willingness to use device for long term. These will be reported using descriptive methods for each device, likely as proportions according to the following response options: strongly disagree, disagree, neither agree nor disagree, agree and strongly agree.

CONTACTS AND LOCATIONS:
Overall Officials: Ajay K Gupta, Principal Investigator — Queen Mary University of London
Locations (1):
- Ajay K Gupta, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Anonymized data may be provided after publication of findings on reasonable request as per unit's policy.

REFERENCES:
- [Background] Zhou B, Perel P, Mensah GA, Ezzati M. Global epidemiology, health burden and effective interventions for elevated blood pressure and hypertension. Nat Rev Cardiol. 2021 Nov;18(11):785-802. doi: 10.1038/s41569-021-00559-8. Epub 2021 May 28. PMID 34050340
- [Background] Hypertension in adults: diagnosis and management. London: National Institute for Health and Care Excellence (NICE); 2023 Nov 21. Available from http://www.ncbi.nlm.nih.gov/books/NBK547161/ PMID 31577399
- [Background] Muntner P, Shimbo D, Carey RM, Charleston JB, Gaillard T, Misra S, Myers MG, Ogedegbe G, Schwartz JE, Townsend RR, Urbina EM, Viera AJ, White WB, Wright JT Jr. Measurement of Blood Pressure in Humans: A Scientific Statement From the American Heart Association. Hypertension. 2019 May;73(5):e35-e66. doi: 10.1161/HYP.0000000000000087. PMID 30827125
- [Background] de la Sierra A, Gorostidi M, Banegas JR, Segura J, de la Cruz JJ, Ruilope LM. Nocturnal hypertension or nondipping: which is better associated with the cardiovascular risk profile? Am J Hypertens. 2014 May;27(5):680-7. doi: 10.1093/ajh/hpt175. Epub 2013 Sep 23. PMID 24061070
- [Background] Townsend RR. Out-of-Office Blood Pressure Monitoring: A Comparison of Ambulatory Blood Pressure Monitoring and Home (Self) Monitoring Of Blood Pressure. Hypertension. 2020 Dec;76(6):1667-1673. doi: 10.1161/HYPERTENSIONAHA.120.14650. Epub 2020 Oct 5. No abstract available. PMID 33012202
- [Background] Stergiou GS, Mukkamala R, Avolio A, Kyriakoulis KG, Mieke S, Murray A, Parati G, Schutte AE, Sharman JE, Asmar R, McManus RJ, Asayama K, De La Sierra A, Head G, Kario K, Kollias A, Myers M, Niiranen T, Ohkubo T, Wang J, Wuerzner G, O'Brien E, Kreutz R, Palatini P; European Society of Hypertension Working Group on Blood Pressure Monitoring and Cardiovascular Variability. Cuffless blood pressure measuring devices: review and statement by the European Society of Hypertension Working Group on Blood Pressure Monitoring and Cardiovascular Variability. J Hypertens. 2022 Aug 1;40(8):1449-1460. doi: 10.1097/HJH.0000000000003224. Epub 2022 Jun 16. PMID 35708294
- [Background] Stevens SL, Wood S, Koshiaris C, Law K, Glasziou P, Stevens RJ, McManus RJ. Blood pressure variability and cardiovascular disease: systematic review and meta-analysis. BMJ. 2016 Aug 9;354:i4098. doi: 10.1136/bmj.i4098. PMID 27511067
- [Background] Sola J, Cortes M, Perruchoud D, De Marco B, Lobo MD, Pellaton C, Wuerzner G, Fisher NDL, Shah J. Guidance for the Interpretation of Continual Cuffless Blood Pressure Data for the Diagnosis and Management of Hypertension. Front Med Technol. 2022 May 17;4:899143. doi: 10.3389/fmedt.2022.899143. eCollection 2022. PMID 35655524
- [Background] Islam SMS, Chow CK, Daryabeygikhotbehsara R, Subedi N, Rawstorn J, Tegegne T, Karmakar C, Siddiqui MU, Lambert G, Maddison R. Wearable cuffless blood pressure monitoring devices: a systematic review and meta-analysis. Eur Heart J Digit Health. 2022 May 2;3(2):323-337. doi: 10.1093/ehjdh/ztac021. eCollection 2022 Jun. PMID 36713001
- [Background] Tan I, Gnanenthiran SR, Chan J, Kyriakoulis KG, Schlaich MP, Rodgers A, Stergiou GS, Schutte AE. Evaluation of the ability of a commercially available cuffless wearable device to track blood pressure changes. J Hypertens. 2023 Jun 1;41(6):1003-1010. doi: 10.1097/HJH.0000000000003428. Epub 2023 Apr 3. PMID 37016925
- [Background] Hu JR, Martin G, Iyengar S, Kovell LC, Plante TB, Helmond NV, Dart RA, Brady TM, Turkson-Ocran RN, Juraschek SP. Validating cuffless continuous blood pressure monitoring devices. Cardiovasc Digit Health J. 2023 Jan 16;4(1):9-20. doi: 10.1016/j.cvdhj.2023.01.001. eCollection 2023 Feb. PMID 36865583
- [Background] Chow CK, Teo KK, Rangarajan S, Islam S, Gupta R, Avezum A, Bahonar A, Chifamba J, Dagenais G, Diaz R, Kazmi K, Lanas F, Wei L, Lopez-Jaramillo P, Fanghong L, Ismail NH, Puoane T, Rosengren A, Szuba A, Temizhan A, Wielgosz A, Yusuf R, Yusufali A, McKee M, Liu L, Mony P, Yusuf S; PURE (Prospective Urban Rural Epidemiology) Study investigators. Prevalence, awareness, treatment, and control of hypertension in rural and urban communities in high-, middle-, and low-income countries. JAMA. 2013 Sep 4;310(9):959-68. doi: 10.1001/jama.2013.184182. PMID 24002282
- [Background] Beaney T, Schutte AE, Stergiou GS, Borghi C, Burger D, Charchar F, Cro S, Diaz A, Damasceno A, Espeche W, Jose AP, Khan N, Kokubo Y, Maheshwari A, Marin MJ, More A, Neupane D, Nilsson P, Patil M, Prabhakaran D, Ramirez A, Rodriguez P, Schlaich M, Steckelings UM, Tomaszewski M, Unger T, Wainford R, Wang J, Williams B, Poulter NR; MMM Investigators*. May Measurement Month 2019: The Global Blood Pressure Screening Campaign of the International Society of Hypertension. Hypertension. 2020 Aug;76(2):333-341. doi: 10.1161/HYPERTENSIONAHA.120.14874. Epub 2020 May 18. PMID 32419505
- [Background] Sola J, Vybornova A, Fallet S, Polychronopoulou E, Wurzner-Ghajarzadeh A, Wuerzner G. Validation of the optical Aktiia bracelet in different body positions for the persistent monitoring of blood pressure. Sci Rep. 2021 Oct 19;11(1):20644. doi: 10.1038/s41598-021-99294-w. PMID 34667230
- [Background] Komori T, Eguchi K, Hoshide S, Williams B, Kario K. Comparison of wrist-type and arm-type 24-h blood pressure monitoring devices for ambulatory use. Blood Press Monit. 2013 Feb;18(1):57-62. doi: 10.1097/MBP.0b013e32835d124f. PMID 23263536
- [Background] International Organization for Standardization, Non-invasive sphygmomanometers - Part 2: Clinical investigation of automated measurement type. 2013.